CLINICAL TRIAL: NCT04563234
Title: Perioperative Cognitive Flexibility Training for the Prevention of Persistent Pain After Thoracic Surgery
Brief Title: Perioperative Cognitive Training in Thoracic Surgery
Acronym: COFLEX-T
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial not funded.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 202007033
Record Dates: First submitted 2020-09-19; First posted 2020-09-24 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Pain, Postoperative; Cognitive Function Abnormal; Lung Cancer
MeSH Terms: conditions — Pain, Postoperative; Cognition Disorders; Lung Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: All study team members will be blinded to the subject assignment to either intervention (cognitive flexibility training) or control groups (crossword puzzle training), except one coordinator who will monitor participant adherence with the cognitive flexibility training, and send prompts or contact participants to understand barriers to adherence.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COFLEX training (Experimental): Neurocognitive training, delivered via a mobile device app
  Interventions: Behavioral: COFLEX neurocognitive training
- Crossword group (Active Comparator): Access to crossword puzzles via a mobile device app
  Interventions: Behavioral: Crossword puzzles

INTERVENTIONS:
Behavioral: COFLEX neurocognitive training — The COFLEX training group will then be provided with the cognitive training module and participants will be required to complete a targeted 30-minute daily training until the day of surgery, and then after the surgery, for a total of 6 weeks.
  Arms: COFLEX training
Behavioral: Crossword puzzles — The control (crossword puzzles) group will be given a training module, where they can access crossword puzzles on the same platform, and can do puzzles whenever they desire over the 6-week time period.
  Arms: Crossword group

SUMMARY:
More than 30% of patients undergoing thoracic surgical procedures develop persistent post-surgical pain (PPSP), which results in impaired functioning, diminished quality of life, and increased risk of chronic opioid use. The proposed project aims to determine whether a prospective, randomized, controlled study of smartphone-based perioperative cognitive flexibility training will reduce the incidence of PPSP in high-risk individuals undergoing thoracic surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 to 75 undergoing thoracic surgery
* Access to an active email account
* Score <50th percentile on Color Word Matching Stroop Test (CWMST) normalized T-score

Exclusion Criteria:

* Unable to complete cognitive testing
* Color blindness assessed via self-report
* Participants who do not speak or read English

The inclusion criteria for the observational cohort will be the same, with the exception of Score ≥50th percentile on Color Word Matching Stroop Test (CWMST) normalized T-score.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06-30 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
The presence of clinically meaningful persistent post-surgical pain 3 months after surgery | 3 months after surgery
  Participants will be asked about pain at or around their surgical area (dichotomous yes/no answer), and rate the intensity of pain, if present, on 0-10 numerical rating scale, where 0=no pain, and 10=worst imaginable pain. The presence of PPSP will be compared between the intervention arm and the control arm

SECONDARY OUTCOMES:
Brief Pain Inventory pain severity | 1 and 3 months after surgery
  BPI (brief pain inventory) severity score will be compared between the study arms. BPI severity score ranges from 0 (least) to 10 (worst)
Brief Pain Inventory pain interference | 1 and 3 months after surgery
  BPI (brief pain inventory) interference score will be compared between the study arms. BPI interference score ranges from 0 (least) to 10 (worst)
PROMIS Anxiety Score | 3 months after surgery
  PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 7 to 35 with higher scores indicating greater severity of anxiety. The score will be compared between the arms
PROMIS Depression score | 3 months after surgery
  PROMIS® (Patient-Reported Outcomes Measurement Information System) is a set of person-centered measures that evaluates and monitors physical, mental, and social health. Each item on the measure is rated on a 5-point scale (1=never; 2=rarely; 3=sometimes; 4=often; and 5=always) with a range in score from 7 to 35 with higher scores indicating greater severity of depression. The score will be compared between the arms.

CONTACTS AND LOCATIONS:
Overall Officials: Simon Haroutounian, PhD, Principal Investigator — Washington University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kehlet H, Jensen TS, Woolf CJ. Persistent postsurgical pain: risk factors and prevention. Lancet. 2006 May 13;367(9522):1618-25. doi: 10.1016/S0140-6736(06)68700-X. PMID 16698416
- [Background] Schug SA, Lavand'homme P, Barke A, Korwisi B, Rief W, Treede RD; IASP Taskforce for the Classification of Chronic Pain. The IASP classification of chronic pain for ICD-11: chronic postsurgical or posttraumatic pain. Pain. 2019 Jan;160(1):45-52. doi: 10.1097/j.pain.0000000000001413. PMID 30586070
- [Background] Smith BH, Torrance N. Epidemiology of neuropathic pain and its impact on quality of life. Curr Pain Headache Rep. 2012 Jun;16(3):191-8. doi: 10.1007/s11916-012-0256-0. PMID 22395856
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu